CLINICAL TRIAL: NCT04552808
Title: To Evaluate the Pharmacokinetics and Safety of Yimitasvir Phosphate Capsules in Subjects With Moderate and Severe Liver Function Impairment and Healthy Subjects in a Single-center, Non-randomized, Open, Single-dose Administration
Brief Title: To Evaluate the Pharmacokinetics and Safety of Yimitasvir Phosphate Capsules in Subjects With Moderate and Severe Liver Function Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DDAG181PA-18-004
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2020-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — yimitasvir

STUDY DESIGN:
Intervention Model Description: This study is divided into four cohorts: healthy subjects in cohort A and C, moderate liver function impairment subjects in cohort B, and severe liver function impairment subjects in cohort D. Cohorts A and B, C and D should be matched in terms of gender, age, and body mass index (BMI).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yimitasvir Phosphate Capsules (Experimental): The mechanism of action of Yimitasvir is the specific inhibition of HCV non-structural protein NS5A
  Interventions: Drug: Yimitasvir Phosphate

INTERVENTIONS:
Drug: Yimitasvir Phosphate — Cohort A: On the first day, 100 mg of Yimitasvir phosphate was given in a single dose on fasted by each subjects
Drug: Yimitasvir Phosphate — Cohort B: were subjects with moderate liver function impairment. On the first day, 100 mg of Yimitasvir phosphate was given in a single dose on fasted by each subjects.
Drug: Yimitasvir Phosphate — Cohort C: Cohort C are healthy subjects, cohorts C and D, should be matched in terms of sex, age, and body mass index (BMI). On the first day, 100 mg of Yimitasvir phosphate was given in a single dose on fasted by each subjects.
Drug: Yimitasvir Phosphate — Cohort D: were subjects with severe liver function impairment. On the first day, 100 mg of Yimitasvir phosphate was given in a single dose on fasted by each subjects.

SUMMARY:
To evaluate the pharmacokinetics and safety of Yimitasvir phosphate capsules in subjects with moderate and severe liver function impairment and healthy subjects in a single-center, non-randomized, open, single-dose administration

DETAILED DESCRIPTION:
A phase I, a single-center, non-randomized, open, single-dose administration study to explore the safety, pharmacokinetics of Yimitasvir phosphate capsules in subjects with moderate and severe liver function impairment and healthy subjects

This study is divided into four cohorts, cohort A and cohort C in healthy subjects, cohort B for moderate liver function impairment participants, cohort D for severe liver function impairment, participants in cohort A and cohort B, group C and group D should be matched in terms of sex, age, and body mass index (BMI). A total of 32 subjects, 8 in each cohort, both male and female, are planned to be enrolled. If a complete PK blood sample is not collected due to subjects' early withdrawal from the study, new subjects will be enrolled to meet the pharmacokinetic parameters that can be evaluated for each cohort of 8 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. subjects and must be 18 to 70 years of age inclusive.
3. Subjects (including partners) have no pregnancy plan within 3 months after the last dose of study drug and voluntarily take effective contraceptive measures.

The following inclusion criteria are only applicable to healthy subjects with normal liver function (cohorts A and C) :

1. The gender and age (±5 years) of subjects in cohort A and C were paired with subjects in cohort B and D, respectively.
2. Body mass index (BMI) : 18-30 kg/m^2 (including critical value) [BMI= weight (kg)/height^2 (m^2)] (BMI matching ±15% with liver dysfunction cohort);
3. Physical examination and vital signs without clinically significant abnormalities.

The following inclusion criteria are only applicable to subjects with liver dysfunction (cohort B and D) :

1. Body mass index (BMI) between 18 and 28 kg/m^2 (including critical value) is allowed for subjects with liver insufficiency without ascites or subjects with subclinical ascites detected only by ultrasound or other imaging.Subjects with clinically significant ascites with liver dysfunction were allowed to have a BMI of 18~30 kg/m^2 (including a threshold).
2. During screening, the severity of patients with liver dysfunction was evaluated according to the Child-Pugh classification : (B/moderate: Child-Pugh score 7~9; Grade C/Severe: Child Pugh score 10~15 points).
3. The liver function status of the subjects was determined to be stable between 1 month before taking the experimental drug and the end of the study, with no significant change.

Exclusion Criteria:

1. Use of >5 cigarettes per day during the past 3 months.
2. Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies).
3. History of alcohol abuse .
4. Donation or loss of blood over 400 mL within 3 months prior to screening. 5.12-lead ECG with clinically significant.

The following exclusion criteria apply only to healthy subjects with normal liver function (cohorts A and C) :

1. Hepatitis B surface antigen (HBsAg) was screened for positivity.
2. Have taken any drug (including prescription and non-prescription drugs, herbal preparations) within 2 weeks prior to taking the experimental drug.

The following exclusion criteria apply only to subjects with liver function impairment (cohorts B and D) :

1. ALT>10×ULN；
2. Absolute count of neutrophils <0.75×10^9/L;
3. PLT<50×10^9/L
4. HGB<60 g/L
5. AFP >100 ng/mL; If 20 ng/mL≤AFP≤100 ng/mL, liver ultrasound examination or other imaging examinations (CT, MRI, etc.) are required to exclude subjects with suspected HCC.
6. eGFR<60 mL/min/1.73m^2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From Days 1-7
  Incidence of adverse events
Cmax | From Days 1-5
  Maximum plasma concentration of study drugs
AUC | From Days 1-5
  Maximum plasma concentration of study drugs

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China